CLINICAL TRIAL: NCT07004829
Title: Efficacy of a Mobile Chat-based Exercise Counselling Intervention (ChatEx) for Increasing and Maintaining Exercise Behaviour in Older Cancer Survivors: A Randomized Controlled Trial
Brief Title: Exercise Counseling Via Mobile Chat for Older Cancer Survivors
Acronym: ChatEx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22233291
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Survivorship; Elderly; Exercise
Keywords: Cancer survivors; Exercise counselling; Instant messaging
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent randomizer will prepare a computer-generated list of random assignments in sealed, sequentially numbered opaque envelopes. Permuted blocks of different sizes will be used to aid allocation concealment. A secure copy of the randomization list will be kept by independent personnel, serving as a central allocation centre. The outcome assessors and statistician performing data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChatEx (Experimental): The ChatEx intervention aims to increase exercise behavior in older cancer survivors through 12 weeks of mobile messages delivered by a trained counselor, complemented by two face-to-face sessions at weeks 1 and 6 to enhance effectiveness and minimize costs. Participants will personalize their message delivery preferences (application, timing, format, language style) from a pre-existing library of text, audio, images, videos, and stickers. Messages, structured using the M-PAC framework, will provide factual information and initiate conversations, with the counselor offering real-time replies to encourage participants to meet exercise guidelines (≥150 minutes of moderate aerobic and two resistance exercise sessions per week).
  Interventions: Behavioral: Exercise counselling via instant messaging
- Control (No Intervention): The control group participants will receive a one-page written information sheet on the recommended exercise guidelines and exercise safety precautions in cancer survivors. Also, they will receive 3-4 messages via IM monthly on non-exercise-related self-management tips of cancer survivorship. They can receive the ChatEx intervention upon completion of the study.

INTERVENTIONS:
Behavioral: Exercise counselling via instant messaging — The 12 weeks of messages will be sent by a trained counsellor. At baseline, participants will select their desired IM application (WhatsApp/WeChat), timing of messages (morning/noon/afternoon), message format (audio/text), and language style (spoken/written). The message library, established in the HMRF-funded study, consists of messages in text and pre-recorded voice message formats, images, videos, and stickers. Each week starts with messages on factual information and ends with a question to initiate conversations to clear any queries; counsellor will provide real-time replies. The 12-week messages are structured based on the M-PAC framework.
  Arms: ChatEx

SUMMARY:
The objective of the study is to determine the efficacy of a 12-week mobile chat-based exercise counselling intervention (ChatEx) for increasing exercise behaviour (operationalized as self-reported aerobic MVPA) at 3-month (primary analysis, post-intervention) and 6-month (3-month post-intervention) among older cancer survivors. This will be a randomized controlled, assessor-blind trial conforming to the CONSORT guidelines. A total of 196 cancer survivors aged over 60 who have completed curative treatment and screened as having an ECOG performance status of 0 or 1 will be recruited and randomized into intervention and control groups. It is expected that upon intervention completion, the intervention group will exhibit increased and sustained exercise behaviors compared to the control group. Study instruments will be Physical Activity Scale for the Elderly, 6-minute walk test, grip strength, Edmonton Frail Scale, European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire, M-PAC constructs, and a background questionnaire. The intervention comprises of 12 weeks of messages aimed at promoting physical activity structured with the multi-process action control framework complemented with two face-to-face exercise instructional sessions at week 1 and week 6. The control group participants will receive a one-page written information sheet on the recommended exercise guidelines and exercise safety precautions in cancer survivors. Also, they will receive 3-4 messages via IM monthly on non-exercise-related self-management tips of cancer survivorship. They can receive the ChatEx intervention upon completion of the study. Intention-to-treat analysis will be performed.

DETAILED DESCRIPTION:
Older adults account for more than half of cancer diagnoses. With advances in detection and treatment, older adults constitute the fastest-growing segment in the cancer population. A history of cancer has been found to increase the odds of and accelerate functional decline, suggesting that cancer and/or its treatment alters aging trajectories. Therapeutic interventions are therefore needed to mitigate the consequences of cancer and aging. Robust evidence indicates that exercise attenuates the major hallmarks of aging. Meanwhile, exercise is recommended by multiple best practice guidelines to alleviate the adverse sequelae of cancer. Well-documented benefits include improvements in physical functioning and quality of life (QoL), reduction of cancer-related symptoms (e.g., fatigue, insomnia, depression), and decreasing risk of recurrence, secondary cancers, and mortality.

Exercise counseling, which involves advice and discussions to promote exercise, is a less intensive and more scalable approach than supervised exercise sessions. Instant messaging (IM) offers a promising platform for delivering exercise counseling due to its accessibility, customizability, and widespread use. This study utilizes the Multi-Process Action Control (M-PAC) framework, which emphasizes reflective, regulatory, and reflexive processes to overcome barriers to exercise adherence. The study hypothesizes that ChatEx, an IM-based exercise counseling intervention grounded in the M-PAC framework, will be effective in increasing and maintaining exercise behavior among older cancer survivors.

This study aims to evaluate the efficacy of a 12-week mobile chat-based exercise counseling intervention (ChatEx) for increasing exercise behavior in older cancer survivors. The primary objective is to determine if ChatEx can increase exercise behavior at both 3-month (post-intervention) and 6-month (3-month post-intervention) time points. Secondary aims include examining the intervention's impact on other exercise parameters, exercise capacity, grip strength, frailty, and quality of life, as well as exploring the mediating roles of Multi-Process Action Control (M-PAC) constructs and participant engagement in changing exercise behavior.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥60
2. diagnosed with stage I-III non-metastatic cancer (rationale: exercise levels and interests in receiving exercise interventions are similar across cancer types in post-treatment survivors
3. completed primary treatment with curative intent (rationale: post-cancer treatment period imposes less exercise barriers related to treatment schedule and side-effects, and is most desired by cancer patients to start/resume exercising
4. can communicate in Cantonese or Mandarin
5. have an ECOG performance status of 0 or 1
6. own a smartphone and proficient in using IM

Exclusion Criteria:

1. contraindications to unsupervised exercise (e.g., dementia, recent myocardial infarction or stroke, chronic obstructive pulmonary disease, walker or wheelchair use)
2. already performing ≥150 minutes of moderate or 75 minutes of vigorous aerobic exercise and two sessions of resistance exercise per week (already meeting recommended exercise guidelines).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Exercise behaviour | (a) pre-intervention at study entry (T0, baseline); (b) 3-month (T1; post-intervention); (c) 6-month (T2; 3 months post-intervention)
  Exercise behaviour (primary outcome) is operationalized as the self-reported time spent in aerobic MVPA per week. It will be assessed using the Physical Activity Scale for the Elderly (PASE) [35], a 12-item scale on three components of physical activity of older adults, including leisure-time activity (light/moderate/vigorous aerobic exercise and resistance exercise), household activity, and work-related activity. The number of hours spent on each activity/day over a 7-day period is recorded. Frequency is multiplied by duration to obtain the total time spent in aerobic MVPA. The total time spent in resistance exercise will be extracted in the same manner. An overall PASE score will be calculated to estimate total exercise time (all types of activities) by summing all components according to the item weights specified. Besides, objectively-measured time spent in MVPA will be measured by instructing participants to wear an activity sensor for 2 consecutive days at each time point.

SECONDARY OUTCOMES:
Exercise capacity | (a) pre-intervention at study entry (T0, baseline); (b) 3-month (T1; post-intervention); (c) 6-month (T2; 3 months post-intervention)
  Exercise capacity will be measured by the 6-minute walk test, which is well-correlated with peak VO2 and highly reproducible. Participants will be instructed to walk at their fastest pace and cover the longest possible distance in 6 minutes.
Grip strength | (a) pre-intervention at study entry (T0, baseline); (b) 3-month (T1; post-intervention); (c) 6-month (T2; 3 months post-intervention)
  Grip strength will be assessed using a dynamometer for six attempts in an alternating bilateral sequence (three with each arm, with a rest period of 30s between each trial). An average of the attempts will be recorded.
Health-related quality of life | (a) pre-intervention at study entry (T0, baseline); (b) 3-month (T1; post-intervention); (c) 6-month (T2; 3 months post-intervention)
  Health-related quality of life will be measured using the 30-item European Organization for research and Treatment of Cancer Core Quality of Life Questionnaire, which has been validated in Chinese cancer patients with satisfactory reliability
Frailty | (a) pre-intervention at study entry (T0, baseline); (b) 3-month (T1; post-intervention); (c) 6-month (T2; 3 months post-intervention)
  Frailty will be measured using the 11-item Edmonton Frail Scale. This covers nine domains of frailty (e.g., cognition, mood, functional performance). Higher total scores represent more severe frailty states.
M-PAC constructs | (a) pre-intervention at study entry (T0, baseline); (b) 3-month (T1; post-intervention); (c) 6-month (T2; 3 months post-intervention)
  M-PAC constructs (e.g., affective attitude, instrumental attitude, perceived capability, perceived opportunity, habit, identity) will be measured using 21 items designed by our co-A (Rhodes, M-PAC founder).

CONTACTS AND LOCATIONS:
Overall Officials: Denise Shuk Ting Cheung, Ph.D., Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request as decided by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 3 years after the manuscript on main findings is published.